CLINICAL TRIAL: NCT00310128
Title: Phase II Study of Induction Therapy Comprising Etoposide, Methylprednisolone, Cytarabine, and Cisplatin (ESHAP) Followed by Consolidation Therapy Comprising Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan in Patients With Relapsed or Refractory AIDS-Related Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Followed by Rituximab and Yttrium Y 90 Ibritumomab Tiuxetan in Treating Patients With Relapsed or Refractory AIDS-Related Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply unavailable
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AMC-044; CDR0000467797 (Other: NCI)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: AIDS-related Lymphoma; Adult Non-Hodgkin's Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related immunoblastic large cell lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult Burkitt's lymphoma; noncontiguous stage II adult Burkitt's lymphoma; recurrent adult Burkitt's lymphoma; stage I adult Burkitt's lymphoma; stage III adult Burkitt's lymphoma; stage IV adult Burkitt's lymphoma; anaplastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma, AIDS-Related; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Follicular; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Cisplatin; Cytarabine; Etoposide; Methylprednisolone; Rituximab; ibritumomab tiuxetan; Immunization, Passive; Biological Therapy; Drug Therapy; Antibodies, Monoclonal; Radiotherapy; Radioimmunotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: cytarabine
Drug: etoposide
Drug: methylprednisolone
Drug: rituximab
Drug: yttrium Y 90 ibritumomab tiuxetan
Procedure: antibody therapy
Procedure: biological therapy
Procedure: chemotherapy
Procedure: monoclonal antibody therapy
Procedure: radiation therapy
Procedure: radioimmunotherapy
Procedure: radioisotope therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as etoposide, methylprednisolone, cytarabine, and cisplatin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab and yttrium Y 90 ibritumomab tiuxetan, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them without harming normal cells. Giving more than one drug (combination chemotherapy) together with rituximab and yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with rituximab and yttrium Y 90 ibritumomab tiuxetan works in treating patients with relapsed or refractory AIDS-related non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall survival rate at one year in patients with relapsed or refractory AIDS-related non-Hodgkin's lymphoma treated with consolidation therapy comprising rituximab and yttrium Y 90 ibritumomab tiuxetan (radioimmunotherapy) given after induction therapy comprising etoposide, methylprednisolone, cytarabine, and cisplatin (ESHAP).
* Describe the toxicity profile of radioimmunotherapy as consolidation therapy, including changes in immunologic and virologic parameters over time, in these patients.
* Determine the overall disease-free survival of patients receiving ESHAP as induction therapy followed by radioimmunotherapy as consolidation therapy.

Secondary

* Determine the effect of ESHAP as induction therapy and radioimmunotherapy as consolidation therapy on HIV-1 viral load, CD4 and CD8 cells, and quantitative immunoglobulin levels in patients on concurrent highly active antiretroviral therapy (HAART).
* Determine the objective response rates (complete and partial response) in patients treated with this regimen.
* Determine the toxicity of ESHAP as induction therapy in these patients.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive ESHAP chemotherapy comprising etoposide IV over 2 hours on days 1-4, methylprednisolone IV over 15-30 minutes on days 1-5, cisplatin IV continuously over 96 hours on days 1-4, and cytarabine IV over 2 hours on day 5. Treatment repeats every 21-28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Approximately 21-52 days after completion of ESHAP chemotherapy, patients proceed to consolidation therapy.
* Consolidation therapy: Patients receive radioimmunotherapy comprising rituximab IV over 3-4 hours followed by indium In 111 ibritumomab tiuxetan (for radioimaging) IV over 10 minutes on day 1. Patients then undergo imaging on days 1 and 2. If biodistribution is acceptable, patients receive rituximab IV over 3-4 hours followed by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.

After completing study treatment, patients are followed every 2 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically documented B-cell non-Hodgkin's lymphoma, including any of the following histologic types:
* Follicular large B-cell lymphoma (follicular, grade 3)
* Follicular mixed cell lymphoma (follicular, grade 2)
* Diffuse mixed cell lymphoma
* Diffuse large B-cell lymphoma
* Immunoblastic lymphoma
* Burkitt or Burkitt-like lymphoma
* Anaplastic large cell lymphoma
* Primary effusion lymphoma
* All stages eligible
* Seropositive for HIV by any approved test or positive HIV-1 RNA in plasma at anytime in the past
* Prior documentation of HIV seropositivity allowed
* Received 1 prior anthracycline-based regimen of curative intent
* No more than 1 prior regimen
* Measurable or evaluable disease
* Evaluable disease defined as not having bidimensional measurements (i.e., gastric or marrow involvement) but can be followed for response by other diagnostic tests, such as gallium scan, positron emission tomography (PET) imaging and/or bone marrow biopsy
* No primary CNS lymphoma
* Lymphomatous meningitis or brain metastasis eligible provided other measurable systemic lymphomatous disease is also present
* Less than 25% bone marrow involvement with lymphoma
* Concurrent effective highly active anti-retroviral therapy (HAART) required at study entry
* HIV viral load < 100,000 copies/mL if HAART was not used previously

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Bilirubin ≤ 2.0 mg/dL (unless elevated due to lymphomatous involvement of the liver or biliary tract OR due to other HIV medications [e.g., indinavir or atazanavir])
* Creatinine < 2.0 mg/dL (< 2.6 mg/dL if due to use of tenofovir or truvada) OR creatinine clearance ≥ 60 mL/min
* Granulocyte count > 1,000/mm^3 (unless abnormal due to lymphomatous involvement of the bone marrow)
* Platelet count > 75,000/mm^3 (unless abnormal due to lymphomatous involvement of the bone marrow or HIV-related thrombocytopenia)
* No acute intercurrent infection that may interfere with study participation
* Mycobacterium avium allowed
* No second active tumor except nonmelanomatous skin cancer, carcinoma in situ of the cervix, or Kaposi's sarcoma not requiring systemic chemotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* No serious, ongoing nonmalignant disease or infection that would compromise study objectives
* No antimurine antibody (HAMA) reactivity
* No history of any cutaneous or mucocutaneous reaction from prior rituximab administration
* No history of cutaneous or mucocutaneous reactions or diseases severe enough to cause hospitalization or an inability to eat for ≥ 2 days

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Fully recovered from all toxicities associated with prior surgery, radiotherapy, chemotherapy, or immunotherapy
* Prior chronic therapy with potentially myelosuppressive agents allowed provided hematologic criteria are met at study entry
* No radiotherapy within the past 4 weeks, unless for emergency conditions secondary to lymphoma (i.e., cord compression)
* No anticancer therapy within the past 3 weeks (6 weeks for nitrosourea or mitomycin C)
* No rituximab within 6 weeks before study radioimmunotherapy
* No investigational agent(s) within the past 4 weeks, unless these are antiretroviral agents available on a compassionate use basis
* No prior external beam radiotherapy to > 25% of active bone marrow (involved field or regional)
* No major surgery, other than diagnostic surgery, within the past 4 weeks
* No prior myeloablative therapies with autologous bone marrow transplantation, peripheral blood stem cell rescue, or failed stem cell collection
* No prior radioimmunotherapy
* No pegfilgrastim within 4 weeks before study radioimmunotherapy
* No other growth factors within 2 weeks before and after study radioimmunotherapy
* No other concurrent myelosuppressive antineoplastic agents after receipt of study radioimmunotherapy until blood counts recover
* No zidovudine-containing regimens (including lamivudine and trizivir) during and for ≥ 2 months after completion of study radioimmunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M. Levine, MD, Study Chair — University of Southern California; Anil Tulpule, MD — University of Southern California